CLINICAL TRIAL: NCT06690021
Title: Comparing the Effect of Adding Dexmedetomidine to Bupivacaine in Classical and Modified Thoracolumbar Interfascial Plane Block on Postoperative Pain in Patients Undergoing Lumbar Disc Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohand Mohamed Fathy Salem, resident doctor anesthesia, Intensive Care and Pain Management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexmedetomidine TLIP lumbar
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Disc Surgery
Keywords: Dexmedetomidine; Classical and Modified Thoracolumbar Interfascial Plane Block
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent anesthesiologist randomly using computer-generated random numbers divided the patients into 2 groups :(Group 1 and Group 2). Each group will include 15 patients. We discreetly placed the randomization results in envelopes until the end of the study. The researchers who were responsible for postoperative follow-up and data processing were blinded to the group allocation during the whole study period. All patients were also blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): Classical Thoracolumbar Interfascial Plane Block
  Interventions: Drug: Dexmedetomidine
- group 2 (Experimental): Modified Thoracolumbar Interfascial Plane Block
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Thoracolumbar Interfascial Plane Block using Bupivacaine and dexmedetomidine

SUMMARY:
Spinal surgeries are frequently conducted to stabilize the vertebrae and discs of the spine. These surgeries typically require substantial manipulation of subcutaneous tissues, bones, and ligaments . Postoperative pain relates to mechanical irritation, compression, and postoperative inflammation. The uncontrolled pain could promote the development of chronic persistent pain and worsen independence, mood, and quality of life. Effective pain management facilitates early mobilisation and accelerates hospital discharge. this study aim to investigate the effectiveness of a mixture of dexmedetomidine and bupivacaine in classical thoracolumbar interfascial plane block compare to modified thoracolumbar interfascial plane block on postoperative pain in patients undergoing lumbar disc surgeries.

DETAILED DESCRIPTION:
Postoperative pain control after spinal surgeries has been a topic of interest for researchers in the past decade. Indeed, poor pain control can not only impact patient satisfaction but also delay rehabilitation and increase healthcare costs.

The thoracolumbar interfascial plane (TLIP) block was defined by Hand et al. for reducing pain following spinal surgery. In this block, the anesthetic drug is administered between the multifidus and longissimus muscles to target the dorsal ramus of the thoracolumbar nerves. The TLIP block was later modified by Ahiskalioglu et al., with the involvement of the administration of a local anesthetic between the longissimus and iliocostalis, which was observed to demonstrate a dermatomal dispersion similar to that by the TLIP block.

Dexmedetomidine is highly specific and highly selective a2-adrenoceptive agonist and it's action is selective to the CNS without the unwanted effect on the CVS that would result from a activation . It has been found that, in many experimental and clinical regional block practices, the addition of dexmedetomidine to the local anesthetic reduces tissue and nerve damage, increases duration of sensory and motor block, and reduces postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years old

  * Both sex
  * Patients who were in risk-scoring groups I-II of the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* • Patient refusal.

  * coagulation disorders that affect the blood's clotting activities e.g.: Hemophilia.
  * skin lesions or infection at site of proposed needle.
  * known allergy to local anesthetics or dexmedetomidine.
  * patients suffering from mental disease as cannot Assess the Visual Analogue Scale (VAS) that measures pain intensity as, mental retardation & psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
total opioid consumption | 24 hours
  To assess the total perioperative (intraoperative and 24 h postoperative) opioid consumption in the first 24 h.

SECONDARY OUTCOMES:
post operative VAS score | 24 hours
  Postoperative pain will be assessed using an 11-point (0=no pain and 10=worst pain) VAS scale. VAS for pain at rest and when coughing will be assessed serially at 1, 2, 4, 8, 16 and 24 h after surgery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ammar MA, Taeimah M. Evaluation of thoracolumbar interfascial plane block for postoperative analgesia after herniated lumbar disc surgery: A randomized clinical trial. Saudi J Anaesth. 2018 Oct-Dec;12(4):559-564. doi: 10.4103/sja.SJA_177_18. PMID 30429737
- [Background] Sarvesh B, Shivaramu BT, Sharma K, Agarwal A. Addition of Dexmedetomidine to Ropivacaine in Subcostal Transversus Abdominis Plane Block Potentiates Postoperative Analgesia among Laparoscopic Cholecystectomy Patients: A Prospective Randomized Controlled Trial. Anesth Essays Res. 2018 Oct-Dec;12(4):809-813. doi: 10.4103/aer.AER_141_18. PMID 30662112
- [Background] Nasr DA, Abdelhamid HM. The efficacy of caudal dexmedetomidine on stress response and postoperative pain in pediatric cardiac surgery. Ann Card Anaesth. 2013 Apr-Jun;16(2):109-14. doi: 10.4103/0971-9784.109744. PMID 23545865
- [Background] Tantri AR, Sukmono RB, Lumban Tobing SDA, Natali C. Comparing the Effect of Classical and Modified Thoracolumbar Interfascial Plane Block on Postoperative Pain and IL-6 Level in Posterior Lumbar Decompression and Stabilization Surgery. Anesth Pain Med. 2022 Apr 12;12(2):e122174. doi: 10.5812/aapm-122174. eCollection 2022 Apr. PMID 36061531
- [Background] Mondal S, Pandey RK, Kumar M, Sharma A, Darlong V, Punj J. Analgesic efficacy of classical thoracolumbar interfascial plane block versus modified thoracolumbar interfascial plane block in patients undergoing lumbar disc surgeries: A comparative, randomised controlled trial. Indian J Anaesth. 2024 Apr;68(4):366-373. doi: 10.4103/ija.ija_1153_23. Epub 2024 Mar 13. PMID 38586260
- [Background] Khan MA, Gupta M, Sharma S, Kasaudhan S. A comparative study of ultrasound assisted versus landmark technique for combined spinal-epidural anaesthesia in patients undergoing lower limb orthopaedic surgery. Indian J Anaesth. 2022 Apr;66(4):272-277. doi: 10.4103/ija.ija_775_21. Epub 2022 Apr 20. PMID 35663223